CLINICAL TRIAL: NCT06568900
Title: A Randomized Controlled Trial to Evaluate the Impact of ZYN Nicotine Pouch Products on Cigarette Usage and Biomarkers of Exposure in Adult Smokers Over a 12-week Period
Brief Title: Randomized Controlled Trial to Evaluate the Impact of ZYN Nicotine Pouch Products on Cigarette Usage and BoExp in Adult Smokers Over a 12-week Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Match AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00070188
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Tobacco Use
Keywords: nicotine; tobacco; nicotine containing products
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (control) continue smoking their usual brand of CC (Active Comparator)
  Interventions: Other: cigarette smoking
- tobacco flavor and unflavored options of ZYN (Active Comparator)
  Interventions: Other: tobacco flavored and unflavored pouch
- unrestricted flavor options of ZYN (Active Comparator)
  Interventions: Other: unrestricted flavor options pouch

INTERVENTIONS:
Other: cigarette smoking — continue smoking usual brand of cigarette
  Arms: (control) continue smoking their usual brand of CC
Other: tobacco flavored and unflavored pouch — provide tobacco flavored and unflavored options of nicotine pouch
  Arms: tobacco flavor and unflavored options of ZYN
Other: unrestricted flavor options pouch — provide unrestricted flavor options of nicotine pouch
  Arms: unrestricted flavor options of ZYN

SUMMARY:
To verify whether unrestricted access to flavored products is likely to lead to greater reductions in combustible cigarette smoking and decreased exposure to smoking related toxicants.

DETAILED DESCRIPTION:
US adult smokers will be randomized into three groups (Group I: (control) continue smoking their usual brand of CC; Group II: provided with tobacco flavor and unflavored options of ZYN; Group III: provide with unrestricted flavor options of ZYN) to evaluate the impact of availability of different ZYN products on cigarette usage patterns and biomarkers of exposure over a 12-week study period, followed by an 6-week extension for some participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult smokers 22 to 65 years of age (inclusive) at screening.
* Smokes an average of at least 10 commercially available cigarettes per day for the last 12 months.
* Interested in switching from combustible cigarettes to nicotine pouch products.

Exclusion Criteria:

* Participants of childbearing potential (CBP) who are breast-feeding or have a positive pregnancy test.
* Participants who currently use nicotine pouches.
* Participants with known heart disease or medical condition that may adversely affect participant safety

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (total NNAL) in urine | Measured from baseline to week 12
  Concentrations of total NNAL measured in urine and expressed as concentration adjusted for creatinine (pg/mg creat).

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Erkkila, PhD, Study Chair — Swedish Match
Locations (1):
- Rose Research Center, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No